CLINICAL TRIAL: NCT07385339
Title: The Effect of a Nursing Intervention Based on the Comfort Communication Model on Pain and Pain Anxiety in Outpatient Burn Patients: A Randomized Controlled Trial
Brief Title: Comfort Communication Model Intervention for Burn Pain and Pain Anxiety
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TABED 2-25 - 1466
Record Dates: First submitted 2026-01-27; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Burn Patients; Pain Management; Nursing Interventions
Keywords: burn patients; dressing change; pain; pain anxiety; Comfort communication model; nursing intervention
MeSH Terms: conditions — Agnosia; Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comfort Communication Model Group (Experimental): Participants will receive routine outpatient burn dressing care plus a structured COMFORT Communication Model-based nursing communication intervention delivered face-to-face by a wound care nurse during three consecutive dressing visits. Each session lasts ~10 minutes and is implemented during the dressing procedure in a quiet, private setting. Session 1 focuses on building trust, explaining steps, checking understanding, and supporting patient control (Connection/Communication; Orientation and opportunity; Relating). Session 2 focuses on emotional expression and supportive openings (Mindful communication; Openings; Family). Session 3 emphasizes personalization, teamwork, and meaning-making (Relating; Team; Mindful communication). Pain and burn-specific pain anxiety are assessed before each dressing and again ~30 minutes after; final assessment occurs after the 3rd visit.
  Interventions: Other: Comfort Communication Model
- Rutin Care Group (No Intervention): Participants will receive routine outpatient burn dressing care only, without the structured COMFORT-based communication sessions. Baseline data are collected at the first visit, and outcomes are assessed on the same schedule as the intervention arm. Pain and burn-specific pain anxiety are evaluated before each dressing and again ~30 minutes after each procedure, with follow-up assessments completed at the third dressing visit.

INTERVENTIONS:
Other: Comfort Communication Model — COMFORT Communication Model-based nursing communication intervention delivered during outpatient burn dressing changes. Participants in the intervention arm receive three consecutive sessions (~10 minutes each) provided face-to-face by a wound care nurse in a quiet, private setting while routine wound care continues. The nurse uses structured communication aligned with COMFORT components across sessions: Session 1 emphasizes Communication/Connection, Orientation and opportunity, and Relating (clear step-by-step explanation, checking understanding, offering options such as pauses/coping strategies, supporting patient control). Session 2 emphasizes Mindful communication, Openings, and Family (exploring prior experience, inviting emotional expression, identifying supportive persons). Session 3 emphasizes Relating, Team, and Meaning/Mindful communication (personalizing support, reflecting on what helped, meaning-making, and facilitating communication with the care team when appropriate). P
  Arms: Comfort Communication Model Group

SUMMARY:
This single-center, randomized controlled trial will evaluate the effect of a nursing intervention based on the COMFORT Communication Model on procedural pain and burn-specific pain anxiety in adult outpatient burn patients undergoing routine dressing changes at the Adult Burn Center Outpatient Unit of Ankara Bilkent City Hospital. Burn dressing changes are frequently perceived as one of the most painful non-surgical procedures, and repeated exposure to wound care may contribute to anticipatory anxiety and stress, potentially creating a reinforcing cycle in which anxiety amplifies pain and pain increases anxiety. In outpatient burn care, effective nurse-patient communication may play a critical role in improving comfort, supporting coping, and enhancing engagement in ongoing treatment.

Eligible participants will be adults aged 18 years and older with second- or third-degree burns who have experienced at least three prior dressing changes, can communicate in Turkish, and have no major hearing or cognitive impairment or comorbid psychiatric/neurological condition that would prevent understanding of the study procedures. Participants who request withdrawal, require hospitalization during follow-up, or miss two consecutive intervention sessions will be withdrawn from the study. The required minimum sample size was estimated as 62 patients (31 per group) based on power analysis (effect size f=0.30; 80% power).

After providing written and verbal informed consent, participants will be randomly assigned (simple randomization using Random Allocation Software) to either the COMFORT-based communication intervention group or the usual care control group. Data will be collected face-to-face in a quiet and private environment during dressing visits. At the initial visit, participants in both groups will complete a sociodemographic and burn-related information form and baseline assessments. Pain intensity will be evaluated using a Verbal Rating Scale and a Numeric Rating Scale, and pain anxiety will be assessed using the Burn-Specific Pain Anxiety Scale; perceived stress will also be measured.

The intervention will be delivered by a wound care nurse during three consecutive dressing sessions. Each session is structured to last approximately 10 minutes and uses specific components of the COMFORT Communication Model tailored to the dressing-change context. In Session 1, the focus is on establishing trust, providing clear information, and supporting patient control through Connection/Communication, Orientation and opportunity, and Relating strategies (e.g., explaining the procedure step-by-step, checking understanding, offering supportive options, and inviting the patient to signal if they want pauses). In Session 2, the focus shifts to creating space for emotions and strengthening supportive openings using Mindful communication, Openings, and Family components (e.g., exploring how the prior session felt, inviting expression of concerns, and identifying supportive persons). In Session 3, communication emphasizes personalization, meaning-making, and teamwork by integrating Relating, Team, and Meaning-focused prompts (e.g., reflecting on what was most helpful, supporting adaptive coping, and, if appropriate, facilitating communication with the clinical team). Throughout all sessions, routine wound care will continue as standard practice in both groups.

Outcomes will be assessed repeatedly across the three dressing sessions. Pain and pain anxiety will be assessed before each dressing, and follow-up assessments will be repeated approximately 30 minutes after the dressing procedure. The primary objective is to determine whether COMFORT model-based nursing communication reduces procedural pain intensity and burn-specific pain anxiety compared with usual care during outpatient dressing changes. A secondary objective is to evaluate whether the intervention reduces perceived stress across sessions. Statistical analyses will include appropriate descriptive and repeated-measures comparisons to examine group differences over time.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years of age or older,
* Patients with at least three dressing experiences
* Patients with 2nd and 3rd degree burns
* No difficulty communicating in Turkish,
* No hearing problems or cognitive impairment,
* No additional mental disorders,
* Willingness to cooperate,
* No additional mental disorders,
* Ability to perform self-care,
* Patients who voluntarily agreed to participate in the study

Exclusion Criteria:

* First-time burn care dressing
* Having a first-degree burn
* Actively receiving inpatient treatment
* Having a neurological or psychiatric condition that prevents reading and understanding data collection tools
* Having difficulty speaking/understanding Turkish

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2026-02-17 (Estimated); Primary Completion 2026-05-08 (Estimated); Study Completion 2026-06-10 (Estimated)

PRIMARY OUTCOMES:
Burn-Specific Pain Anxiety | Baseline (first visit) and across three consecutive dressing sessions (Days 1-3): assessed before each dressing and reassessed ~30 minutes after each dressing; final evaluation after the 3rd session.
  Burn-specific pain anxiety will be measured using the Burn-Specific Pain Anxiety Scale (Turkish version). The scale consists of 8 items scored from 0 ("none") to 10 ("worst imaginable"); total score ranges from 0 to 80, with higher scores indicating greater anxiety related to painful burn care procedures.

SECONDARY OUTCOMES:
Pain Intensity During Dressing Change | Baseline (first visit) and across three consecutive dressing sessions: before each dressing and ~30 minutes after each dressing (Days 1-3).
  Pain intensity will be assessed using two single-item scales: the Verbal Rating Scale (VRS; 5 categories: mild, discomforting, severe, very severe, unbearable) and the Numeric Rating Scale (NRS; 0-10, where 0=no pain and 10=worst imaginable pain). Pain will be measured before each dressing session and re-assessed approximately 30 minutes after the dressing procedure.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wittenberg-Lyles, E., Goldsmith, J., Ragan, S. ve Sanchez-Reilly, S. (2010). Dying with comfort: family illness narratives and early palliative care. Cresskill, NJ: Hampton Press.
- [Background] Wittenberg-Lyles, E., Goldsmith, J. ve Ragan, S.L. (2010). The COMFORT initiative. J Hosp Palliat Nurs. 12(5), 282-292. https://doi.org/10.1097/ NJH.0b013e3181ebb45e
- [Background] Wittenberg E, Ferrell B, Goldsmith J, Ragan SL, Paice J. Assessment of a Statewide Palliative Care Team Training Course: COMFORT Communication for Palliative Care Teams. J Palliat Med. 2016 Jul;19(7):746-52. doi: 10.1089/jpm.2015.0552. Epub 2016 Jun 10. PMID 27285175
- [Background] Tetteh L, Aziato L, Mensah GP, Vehvilainen-Julkunen K, Kwegyir-Afful E. Burns pain management: The role of nurse-patient communication. Burns. 2021 Sep;47(6):1416-1423. doi: 10.1016/j.burns.2020.11.011. Epub 2020 Nov 27. PMID 33277090
- [Background] Goldsmith JV, Wittenberg E, Parnell TA. The COMFORT Communication Model: A Nursing Resource to Advance Health Literacy in Organizations. J Hosp Palliat Nurs. 2020 Jun;22(3):229-237. doi: 10.1097/NJH.0000000000000647. PMID 32282558
- [Background] Davodabady F, Naseri-Salahshour V, Sajadi M, Mohtarami A, Rafiei F. Randomized controlled trial of the foot reflexology on pain and anxiety severity during dressing change in burn patients. Burns. 2021 Feb;47(1):215-221. doi: 10.1016/j.burns.2020.06.035. Epub 2020 Jul 12. PMID 32739224
- [Background] Aghakhani N, Faraji N, Alinejad V, Goli R, Kazemzadeh J. The effect of guided imagery on the quality and severity of pain and pain-related anxiety associated with dressing changes in burn patients: A randomized controlled trial. Burns. 2022 Sep;48(6):1331-1339. doi: 10.1016/j.burns.2021.11.020. Epub 2021 Nov 26. PMID 34924224